CLINICAL TRIAL: NCT00730990
Title: A8801007 A Phase I, Healthy Volunteer Qualification Of Ligand [C 11] PF 04621053 And Randomized Determination Of H3 Receptor Occupancy Of PF 03654746, Using PET
Brief Title: A Phase I, Healthy Volunteer Positron Emission Tomography Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: A8801007
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: Positron Emission Tomography study in healthy volunteers for ligand qualification and receptor occupancy determination.
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; N-ethyl-3-fluoro-3-(3-fluoro-4-(pyrrolidinylmethyl)phenyl)cyclobutanecarboxamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): This arm will have no active treatment.
  Interventions: Other: Positron Emission tomography
- Cohort 2 (Experimental)
  Interventions: Drug: PET Scan with PF-03654746

INTERVENTIONS:
Other: Positron Emission tomography — Positron Emission tomography scans. Part 1of the study : 4 subjects will receive 2 scans a day for 1 day with PET ligand administered in tracer quantities.
  Arms: Cohort 1
Drug: PET Scan with PF-03654746 — If none of the data from Cohort 2 is informative, then: 2) an additional 3 subjects will receive 2 Scans on Day 1 and 1 scan on Day 2 following 3 different doses of PF-03654746. Doses will be determined based upon the outcome of the first intervention.
  Arms: Cohort 2
Drug: PET Scan with PF-03654746 — If none of the data from the previous interventions are informative, then: 3) an additional 3 patients will receive 2 scans on Day 1 and 1 scan on Day 2 following three different doses of PF-0365476. Doses will be determined based upon the outcomes of the previous interventions.
  Arms: Cohort 2
Drug: PET Scan with PF-03654746 — Part 2 of the study will have 3 possible interventions:
  1) 3 subjects in Cohort 2 will receive 2 scans on Day 1 and 1 scan on Day 2 following 3 different doses of PF-03654746 (0.5 mg, 1.5 mg, 4 mg).
  Arms: Cohort 2

SUMMARY:
The primary purpose of this study is to assess central receptor occupancy of PF 03654746 at the H3 receptor after a single oral dose of PF 03654746.

DETAILED DESCRIPTION:
Additional Study Purpose Details: To validate PET ligand which will be used to determine receptor occupancy and to determine receptor occupancy of PF-0367456

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs). A BMI at the lower limit of 17.5 kg/m2 may be rounded up to 18.0 kg/m2; a BMI upper limit of 30.5 kg/m2 may be rounded down to 30.0 kg/m2 and will be acceptable for inclusion.
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* History of febrile illness within 5 days prior to the first dose.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen at Screening or Day 0.
* History of regular alcohol consumption exceeding 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Positive cotinine screen at Screening or Day 0.
* Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study medication (excluding [C-11]PF-04621053).
* 12-lead ECG demonstrating QTc >450 msec at Screening. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued 28 days prior to the first dose of study medication.
* Chronic (every day) use of a histamine (H1, H2) inhibitor(s) within 3 months before screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Overall H3 Receptor Occupancy of PF 03654746. | 48 hours

SECONDARY OUTCOMES:
Binding potential (BP) of [C-11]PF 04621053. | 48 hours
Relationship between serum PF 03654746 concentration and H3 RO (IC50). | 48 hours
H3 RO of PF 03654746 at regions of interest in man | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8801007&StudyName=A%20Phase%20I%2C%20Healthy%20Volunteer%20Positron%20Emission%20Tomography%20Study